CLINICAL TRIAL: NCT04255511
Title: Effects of Orthopedic Mandibular Advancement in Class II Division 1 Malocclusion Children on Pharyngeal Airway and Nocturnal Breathing ; Randomized Controlled Trial
Brief Title: Effects of Orthopedic Mandibular Advancement in Class II Division 1 Malocclusion on Pharyngeal Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mona Montasser, Professor of Orthodontics, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A09061119
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: ClassII Division 1 Malocclusion; Mandibular Retrognathism
MeSH Terms: interventions — Orthodontic Appliances, Fixed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Twin block (Experimental): Removable Functional appliance
  Interventions: Device: Twin Block
- Fixed appliance (Active Comparator): Preadjusted fixed appliance
  Interventions: Device: Fixed orthodontic appliance

INTERVENTIONS:
Device: Twin Block — Functional appliance
  Arms: Twin block
Device: Fixed orthodontic appliance — Braces
  Arms: Fixed appliance

SUMMARY:
This study aims at evaluating the effects of mandibular advancement on pharyngeal airway space and nocturnal breathing in children with skeletal class II division1 malocclusion. Fifty patients will be enrolled in the study divided into control and experimental groups.

DETAILED DESCRIPTION:
The purpose of the present research is not only evaluate the effect of functional appliance on the pharyngeal airway space, but also evaluate its effect on nocturnal breathing of children with skeletal class II.

ELIGIBILITY:
Inclusion Criteria:

1. Skeletal class II division 1 malocclusion due to mandibular retrognathism.
2. Cephalometric angular measurements: SNA ≥ 82, SNB ≤ 78, ANB ≥ 4.
3. Overjet ≥ 6 mm.
4. Patient in circumpubertal stage CVM2 and CVM3.

Exclusion Criteria:

1. History of orthodontic treatment.
2. Presence of craniofacial anomalies or TMJ disorders.
3. Systemic problems that may affect craniofacial growth.
4. Abnormal oral habits.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Pharyngeal airway volume | One year
  CBCT images will be used to measure the pharyngeal airway volume in mm3
Nocturnal breathing | One year
  Pulse oximeter will be used to measure Oxygen Desaturation Index (ODI) and report the number of 3% and/or 4% desaturations.

SECONDARY OUTCOMES:
Maximum expiratory pressure | One year
  Oral expiratory peak flow meter will be used to measure the maximum expiratory pressure as cmH2O.
Craniofacial changes | One year
  Lateral cephalometric images extracted from the CBCT images will be used to measure linear (mm) skeletal, dental and soft tissue changes of maxilla and mandible.
Craniofacial changes | One year
  Lateral cephalometric images extracted from the CBCT images will be used to measure angular (º) skeletal, dental and soft tissue changes of maxilla and mandible.

CONTACTS AND LOCATIONS:
Overall Officials: Mona A Montasser, Phd, Study Chair — Mansoura University; Eman S Radwan, MSc, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Will be based on the facility regulations and approval.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available at the end of the study i.e after 2 years.
Access Criteria: Data will be available through the principle investigator and the study chair.

REFERENCES:
- [Derived] Radwan ES, Maher A, Montasser MA. Effect of functional appliances on sleep-disordered breathing in Class II division 1 malocclusion children: Randomized controlled trial. Orthod Craniofac Res. 2024 Feb;27(1):126-138. doi: 10.1111/ocr.12696. Epub 2023 Jul 31. PMID 37522361